CLINICAL TRIAL: NCT05987137
Title: 2024 National Survey of Early Care and Education (NSECE)
Status: Active, not recruiting | Type: Observational
Sponsor: National Opinion Research Center (Other)
Collaborators: Child Trends (Other); Office of Planning, Research & Evaluation (U.S. Federal Agency); Chapin Hall at the University of Chicago (Other)
Responsible Party: Principal Investigator, Rupa Datta, Distinguished Senior Fellow, National Opinion Research Center
Other Study IDs: HHSP233201500048I-75N98021F003
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Children Under 13
Keywords: Early care and education; Center-based providers; Home-based providers; Caregivers; Child care; Workforce; ECE

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Households: Interviews conducted with the parent or guardian of a child or children under age 13.
  Interventions: Other: No intervention is being administered.
- Home-based providers: Interviews conducted with individuals who provide care in a home-based setting to children under age 13 who are not their own for five or more hours a week.
  Interventions: Other: No intervention is being administered.
- Center-based Providers: Interviews conducted with directors of early care and educations programs that provide care to children not yet in kindergarten.
  Interventions: Other: No intervention is being administered.
- Workforce (Classroom Staff): Interviews conducted with classroom-assigned instructional staff sampled from each center-based provider who completed an interview.
  Interventions: Other: No intervention is being administered.

INTERVENTIONS:
Other: No intervention is being administered. — No intervention is being administered.

SUMMARY:
The National Survey of Early Care and Education (NSECE) captures families' needs, preferences, and choices of non-parental care for children under age 13 and providers' child care and early education offerings. Since the NSECE was last conducted in 2019, the landscape of ECE has changed dramatically. Funding for early childhood programming has grown as policymakers recognize the important role access to ECE plays for families as a work support for parents and an investment in children's future educational and economic opportunities. At the same time, beginning in 2020, the nation experienced the COVID-19 pandemic, leading to significant shifts in the U.S. economy. These circumstances likely altered parents' use of ECE and the labor market and economic forces in which ECE providers operate.

The 2024 NSECE builds on findings from the 2012 and 2019 NSECE to allow for comparisons of supply and demand of child care and early education over the 12 years that span data collection. The 2024 NSECE aims to inform future policy discussions about child care and early education at the local, state, and national levels by providing data to:

* Build on the efforts and lessons from the 2012 and 2019 NSECE to allow for comparisons of child care and early education supply and the early care and education workforce from 2012 to 2024
* Capture the characteristics of households with children under age 13, such as parental employment status and schedules, preferences and choices of non-parental care, and other factors that affect their need for and access to child care and early education
* Document how the field of child care and early education responded to policy initiatives during the period between 2012 and 2024, including changes in supply and demand during the COVID-19 pandemic starting in 2020

DETAILED DESCRIPTION:
In order to create a comprehensive portrait of the availability and use of early care and education, the NSECE is fielding a set of four integrated, nationally representative surveys beginning in 2023. These are surveys of 1) households with children under 13, 2) home-based providers 3) center-based providers, and 4) the center-based provider workforce. Together they characterize the supply of and demand for early care and education in America and permit better understanding of how well families' needs and preferences coordinate with providers' offerings and constraints.

The Household Survey is being conducted with a parent or guardian of a child or children under age 13 in households with at least one member child under age 13. Eligible respondents are identified through the Household Screener based only on the presence of an age-eligible child. Screening is being completed by mail, by phone, by web, and in person. All of these interviews are being conducted by an interviewer, primarily in person. This survey documents the nation's demand for early care and education services. Key questionnaire topics include details on usage of non-parental care, expenditures on non-parental care, parental search behavior for early care and education, and the balance of parental employment with child care needs and availability.

These data will help to answer such research questions as 1) Who is caring for America's children when they are not with their parents and do families with different demographic characteristics have different preferences or different patterns of usage? 2) How do families search for care and how does this vary by age of children, characteristics of parents, location, and availability of licensed slots per population? 3) How and how much do families pay for care? and 4) How many families of different characteristics receive public financial support for ECE, and how does this vary by age of child and type of care utilized?

The Home-based Provider Survey is being conducted with individuals who provide care in a home-based setting for children under age 13 who are not their own for five or more hours a week. Two sample sources contribute providers. One, home-based providers who appear in provider sampling frames constructed from state and national lists were sampled for this survey. These providers are designated as 'listed.' Listed providers are primarily licensed or regulated family day care providers, but also include other formally listed home-based providers such as license-exempt providers or providers participating in Early Head Start. Alternatively, households may be identified as eligible based on their responses to the household screener (specifically, that an adult in the household regularly cares for children not his or her own at least five hours per week in a home-based setting). These providers do not appear in the provider sampling frame and are designated as 'unlisted.' Data collection is being conducted by web, in person, and by telephone with field interviewers.

Key questionnaire topics in the home-based provider questionnaire include enrollment and the characteristics of the children served, rates charged for care, and participation in government programs, household composition, qualifications for and practices regarding early childhood education, use of curricula and activities conducted with children. Portions of the home-based provider questionnaire will contribute to analyses of the ECE workforce and mirror the content of the workforce (classroom staff) questionnaire administered to classroom-assigned instructional staff at center-based providers. Other portions of this questionnaire closely mimic the center-based provider questionnaire (see below), so that enrollment, program participation, provider charges for care, attitudes, orientation and activities data can be accurately compared across all different categories of provider.

These data will answer such questions as 1) What kind of early care and education is available across communities throughout the country? 2) How well does the available supply of early care and education support parents' employment? 3) How do different types of providers vary in their characteristics of care and affordability? and 4) Who are the individuals working in early care and education? What are their experiences in terms of employment characteristics, classroom activities, and professional development? What are their attitudes, practices, and burnout and depression levels?

The inclusion of providers identified through the Household Screener will offer invaluable nationally representative data on family, friend and neighbor providers and is one of the pioneering aspects of the NSECE. Investigators will learn about both paid and unpaid care, including how they differ in their characteristics and their availability to families.

The Center-based Provider Survey will be conducted with directors or administrative staff of ECE programs that provide care to children not yet in kindergarten who were identified from the provider sampling frame built from state or national administrative lists such as state licensing lists, Head Start program records, or pre-K rolls. These providers include regulated, licensed, and other private providers as well. The center-based provider questionnaire is preceded by a Center-based Provider Screener that confirms and updates information from the provider sampling frame and determines eligibility for the center-based provider questionnaire. Topics covered by this instrument include enrollment and characteristics of children served, staffing, prices charged, schedules of service, participation in government programs, and staff compensation and professional development policies. The questionnaire also includes the selection of a representative classroom about which more detailed staffing, compensation, and curriculum information are collected. These data constitute a nationally representative sample of ECE classrooms. This instrument will be administered using web, in-person, and telephone interviewing.

The center-based provider questionnaire data will answer such questions as 1) What kind of early care and education is available across communities throughout the country? 2) How well does the available supply of early care and education support parents' employment? 3) How do different types of providers vary in their characteristics of care and affordability? and 4) How many and what types of providers participate in quality improvement efforts such as staff quality ratings and professional development?

The Workforce (Classroom Staff) Survey sample is comprised of one or two classroom-assigned instructional staff members from each center-based provider who completed a center-based provider interview. Workforce (classroom staff) respondents are drawn from the center-based provider questionnaire data, in which all staff members have been enumerated from a randomly selected classroom. The questionnaire closely mirrors portions of the home-based provider questionnaire, so that the two data sources together can paint a rich portrait of the paid ECE workforce, including center-based and home-based paid providers. (Individuals who are not paid will be profiled as described in the family, friends, and neighbor section above.) Topics include information about the work setting (activities in the classroom, interactions with parents and other staff, availability of professional development and other supports), roles and responsibilities (lead teacher, teacher, assistant teacher, aide), compensation (wages and benefits), and perceived leadership and morale, as well as personal information about qualifications, practices regarding ECE, and burnout, depression, and demographic information.

The workforce (classroom staff) questionnaire is the simplest of the NSECE survey instruments, but these data represent a signal contribution of the study. Before the 2012 study, no nationally representative survey of paid ECE workers had ever been done, yet many of the pressing ECE policy questions require better understanding of ECE workers' qualifications, access to professional development, motivation for working in the field, and nature of participation in the labor market as well as the extent to which paid home-based providers are more generally available for expanding and improving overall ECE supply. Some of the workforce (classroom staff) questionnaire data will allow tabulation by provider program characteristics (such as enrollment size, type of care, geographic location, for-profit/not-for-profit status, and participation in government programs) of factors that have been found in the literature to predict observed quality. These factors include staff qualifications and compensation, use of curricula, availability of professional development, and children's activities while in care. The data will answer such questions as who are the individuals working in early care and education and what are their experiences in terms of employment characteristics, classroom activities, and professional development?

ELIGIBILITY:
Inclusion Criteria:

* Households with at least one child under the age of 13.
* Individuals who care for a child under 13 who are not their own in a home-based setting for at least five hours a week.
* Center-based ECE programs that provide care to children not yet in kindergarten who were identified from the provider sampling frame built from state or national administrative lists such as state licensing lists.
* Respondents for the workforce (classroom staff) survey are selected from the list of instructional staff associated with the randomly selected classroom from the center-based provider interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Households with children under 13 years. Individuals providing at least 5 hours' weekly care to children under 13 years not their own in a home-based setting. Early care and education centers serving children not yet in kindergarten. Individuals working in center-based classrooms.
Sampling Method: Probability Sample
Enrollment: 106200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Need For And Use Of Childcare in Households With Children Under 13 | October 2023 - July 2024
  The household questionnaire collects information on each household's need for and use of early care and education services, including details on usage of non-parental care, expenditures on non-parental care, parental search behavior for early care and education, and the balance of parental employment with child care needs and availability.
Provision And Characteristics Of Child Care Among Center-based Providers | October 2023 - July 2024
  The center-based provider questionnaire collects information on enrollment and characteristics of children served, staffing, prices charged, schedules of service, participation in government programs, and staff compensation and professional development policies. The questionnaire also includes the selection of a representative classroom about which more detailed staffing, compensation, and curriculum information are collected. Individual questionnaire items may be developed into scales by researchers, but specific scales are not prescribed in the study design or analysis plans.
Characteristics And Experiences Of The ECE Workforce | October 2023 - July 2024
  The workforce (classroom staff) questionnaire collects information about the work setting (activities in the classroom, interactions with parents and other staff, availability of professional development and other supports), roles and responsibilities (lead teacher, teacher, assistant teacher, aide), compensation (wages and benefits), and perceived leadership and morale, as well as personal information about qualifications, practices regarding ECE, and burnout, depression, and demographic information. Individual questionnaire items may be developed into scales by researchers, and some standard scales are excerpted in the NSECE questionnaire, but specific scales are not prescribed in the study design or analysis plans.
Provision and characteristics of child care among home-based providers | October 2023 - July 2024
  The workforce (classroom staff) questionnaire collects information about the work setting (activities in the classroom, interactions with parents and other staff, availability of professional development and other supports), roles and responsibilities (lead teacher, teacher, assistant teacher, aide), compensation (wages and benefits), and perceived leadership and morale, as well as personal information about qualifications, practices regarding ECE, and burnout, depression, and demographic information. Individual questionnaire items may be developed into scales by researchers, and some standard scales are excerpted in the NSECE questionnaire, but specific scales are not prescribed in the study design or analysis plans.

CONTACTS AND LOCATIONS:
Overall Officials: Rupa Datta, PhD, Principal Investigator — NORC at the University of Chicago
Locations (1):
- NORC at the University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No